CLINICAL TRIAL: NCT00054613
Title: A Randomized Single-Blind Study of Extracorporeal Photoimmune Therapy With UVADEX in Conjunction With Standard Therapy Alone for the Treatment of Patients With Corticosteroid-Refractory, Corticosteroid-Dependent, or Corticosteroid-Intolerant Chronic Graft-versus-Host Disease
Brief Title: Safety and Efficacy Study of Photopheresis Plus Standard Therapy to Treat Chronic Graft-versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GvHD-SK1
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Graft-versus-Host Disease
Keywords: Graft-versus-Host Disease; Extracorporeal Photopheresis
MeSH Terms: conditions — Graft vs Host Disease | interventions — Methoxsalen; Photopheresis

INTERVENTIONS:
Drug: Methoxsalen
Procedure: Extracorporeal Photopheresis

SUMMARY:
The purpose of this study is to determine whether extracorporeal photoimmune therapy with UVADEX (ECP) added to standard therapy is effective in the treatment of chronic graft-versus-host disease (GvHD).

DETAILED DESCRIPTION:
For patients who survive allogeneic bone marrow transplants greater than 100 days, chronic GvHD is a major cause of non-relapse morbidity and mortality. Depending on the presence of known associated risk factors, chronic GvHD will occur in 20-50% of these transplant recipients, with mortality rates varying from 20 to 70%.

Because a lymphocyte-mediated immune reaction is thought to be involved in GvHD, suppression of these cells by means other than medications could have benefit in the GvHD population.

ECP is a technique in which peripheral white blood cells are exposed to a photoactivatable compound (UVADEX) administered extracorporeally and ultraviolet A light. After cells are reinfused into the patient, their function is altered, thereby activating mechanisms that allow for further regulation of specific lymphocyte populations.

The purpose of this study is to determine whether ECP, in conjunction with standard therapy, is effective in the treatment of chronic GvHD. Efficacy of the therapy with respect to skin manifestations of the disease will be determined by a blinded skin assessor.

ELIGIBILITY:
Inclusion Criteria:

* Documented skin disease classical for chronic GvHD (e.g. hypopigmentation, hyperpigmentation, lichenoid lesions, sclerodermatous lesions)greater than or equal to 100 days post transplantation.
* Patients with documented chronic GvHD that is corticosteroid refractory, corticosteroid dependent or corticosteroid intolerant.
* Women of childbearing potential must agree to use a reliable method of birth control for the duration of this study.
* Patients must weight at least 40 kg (88 lbs.)

Exclusion Criteria:

* Active gastrointestinal bleeding
* Previous treatment with ECP
* Females who are pregnant and/or lactating

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72
Dates: Start 2002-06; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (31):
- United States (11):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Florida, Gainesville, Florida
  - Rush Presbyterian - St. Lukes Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Tufts New England Medical Center, Boston, Massachusetts
  - Brigham and Womens, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Kansas City Cancer Center, Kansas City, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Jewish Hospital, Cincinnati, Ohio
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (4):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Peter MacCallum, East Melbourne
  - Alfred Hospital, Melbourne
  - Royal Melbourne Hospital, Parkville
- General Hospital of Vienna, Vienna, Austria
- France (2):
  - Hopital Edouard Herriot, Lyon
  - Hopital Pitie-Salpetriere, Paris
- Germany (4):
  - University of Dresden, Dresden
  - Universitatis Hautklinik, Essen
  - Universitatsklinikum Leipzig AOR, Leipzig
  - Ludwig-Maximilians-Universitaet Muenchen, München
- Italy (2):
  - Careggi Hospital, Florence
  - San Martino Hospital, Genova
- Instituto Portugues de Oncologia de Francisco Gentil, Lisbon, Portugal
- Klinika hematologie a transfuziologie FN, Bratislava, Slovakia
- Hospital dela Santa Creu i Sant Pau. Universitat Autonoma de Barcelona, Barcelona, Spain
- Kantonsspital Basel, Basel, Switzerland
- Ankara University Medical School, Altındağ, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - Rotherham General Hospital, Rotherham, Yorkshire
  - Glasgow Royal Infirmary, Glasgow

REFERENCES:
- [Background] Smith EP, Sniecinski I, Dagis AC, Parker PM, Snyder DS, Stein AS, Nademanee A, O'Donnell MR, Molina A, Schmidt GM, Stepan DE, Kapoor N, Niland JC, Forman SJ. Extracorporeal photochemotherapy for treatment of drug-resistant graft-vs.-host disease. Biol Blood Marrow Transplant. 1998;4(1):27-37. doi: 10.1016/s1083-8791(98)90007-6. PMID 9701389
- [Background] Greinix HT, Volc-Platzer B, Knobler RM. Extracorporeal photochemotherapy in the treatment of severe graft-versus-host disease. Leuk Lymphoma. 2000 Feb;36(5-6):425-34. doi: 10.3109/10428190009148389. PMID 10784386
- [Derived] Flowers ME, Apperley JF, van Besien K, Elmaagacli A, Grigg A, Reddy V, Bacigalupo A, Kolb HJ, Bouzas L, Michallet M, Prince HM, Knobler R, Parenti D, Gallo J, Greinix HT. A multicenter prospective phase 2 randomized study of extracorporeal photopheresis for treatment of chronic graft-versus-host disease. Blood. 2008 Oct 1;112(7):2667-74. doi: 10.1182/blood-2008-03-141481. Epub 2008 Jul 11. PMID 18621929